CLINICAL TRIAL: NCT06083415
Title: Early Breast Growth in Girls Aged 6 to 8 Years in the Current Environmental Context: Clinical and Biological Parameters, Level of Impregnation With Endocrine Disruptors and Evaluation of the Impact of Environmental Health Measures
Brief Title: Early Breast Growth in Girls Aged 6 to 8 Years in the Current Environmental Context
Acronym: PENELOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RT-17
Record Dates: First submitted 2023-10-04; First posted 2023-10-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Puberty, Precocious; Breast; Environmental Exposure
Keywords: Early puberty; Endocrine disruptors; Girls; Breast growth; Environmental Health Measure
MeSH Terms: conditions — Puberty, Precocious | interventions — Magnetic Resonance Spectroscopy; Hematologic Tests; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 6 to 8 years old girls, presenting with a breast flare-up (Experimental): Girls aged 6 to 8 years old with breast flare (isolated or not) and scheduled for pediatric day hospital stay
  Interventions: Other: Environmental health measures
- 6 to 8 years old girls controls (No Intervention): Girls aged 6 to 8 years old controls, scheduled for pediatric day hospital stay, or an office consultation, or an MRI in radiology

INTERVENTIONS:
Other: Environmental health measures — MRI will be used to confirm the presence of breast buds, to measure the size of the ovaries and uterus, as well as the fraction of fat mass (abdominal, subcutaneous, liver and bone marrow). The bood and urine tests will allow to measure different biological and metabolic parameters. The presence of endocrine disruptors will be determined in the hair. The bone age x ray will be estimate the maturity of the child's skeletal system. Photographs of the teeth will also be taken to be studied by pediatric odontology researchers on the on molar and incisor hypomineralization, known as MIH.
  Other Names: Magnetic Resonance Imaging (MRI); Blood tests; Determination of endocrine disruptors in hair; Urine tests; Bone age x ray; Tooth photography (MIH)
  Arms: 6 to 8 years old girls, presenting with a breast flare-up

SUMMARY:
Various studies show an increase in the number of cases of early puberty in girls with breast development with a variable clinical presentation and evolution. This increasing phenomenon concerns girls between 6 and 8 years old. In a large number of cases, from 70 to 95% depending on the series, no medical cause is found and environmental factors are suspected to be involved.

Descriptive studies of these patients are scarce and not always provide an overview of all the parameters in line with the concept of the exposome.

The PENELOPE clinical trial will allow to analyze a large number of parameters, including the adipose tissue, its metabolism, the endocrine disruptors, and the epigenetic modifications, and to study the impact of environmental health measures in the evolution of these parameters.

The data from the analyses of the endocrine disruptors of the patients will be explored in parallel in experimental models (amphibians, murine, cellular) in order to test potential mechanistic hypotheses.

ELIGIBILITY:
For patients:

Inclusion Criteria:

* Girls aged 6 to 8 years
* Presenting a breast development (isolated or not)
* Undergoing scheduled pediatric day hospital care (HDJ)
* Who agree to participate in the study
* Whose parents agree to their child's participation in the study
* French speaking
* Whose parents speak French
* Affiliated to social security

Exclusion Criteria:

* Organic brain causes of precocious puberty: History of neurocerebral disease (malformations, developmental abnormalities)
* Organic causes of precocious puberty: Mac Cune Albright syndrome, ovarian cyst or tumor and adrenal hyperplasia
* History of chemotherapy or radiation therapy
* Presenting with a communication disorder
* Pregnancy
* Persons under protective measures
* Persons deprived of liberty for judicial or administrative reasons

For controls:

Inclusion Criteria:

* Girls aged 6 to 8
* Tanner stage 1: Absence of breasts and hairiness
* Coming for routine consultation in the pediatric HDJ at Saint-Vincent-de-Paul hospital, or at the BLM practice in Lambersart, or to radiology for an MRI for another medical other medical reason
* Agree to participate in the study
* Whose parents agree to their child's participation in the the study
* French-speaking
* Whose parents speak French
* Affiliated with social security

Exclusion Criteria:

* Signs of puberty (Tanner stages 2, 3, 4 and 5 for breast development) breast development)
* Previous chemotherapy or radiotherapy
* Presenting a communication disorder
* Pregnant women
* Persons under protective supervision
* Persons deprived of their liberty for judicial or administrative reasons

Ages: 6 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Girls aged 6 to 8 years presenting a breast development (isolated or not) or not (controls)
Enrollment: 62 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the size of the breast development measured by Magnetic Resonance Imaging | Baseline, 3 months
  This parameter will allow to describe the clinical evolution of breast development after application of environmental health measures
Change from baseline of the size of ovaries/uterus measured by Magnetic Resonance Imaging | Baseline, 3 months,
  This parameter will allow to describe the clinical evolution of ovaries and uterus after application of environmental health measures
Change from baseline of the abdominal fat surface measured by Magnetic Resonance Imaging | Baseline, 3 months
  This parameter will allow to describe the clinical evolution of the abdominal fat surface after application of environmental health measures
Change from baseline of the weight | Baseline, 3 months, 6 months
  This parameter will allow to describe the clinical evolution of the weight after application of environmental health measures
Change from baseline of the height | Baseline, 3 months, 6 months
  This parameter will allow to describe the clinical evolution of the height after application of environmental health measures
Body mass index (BMI) | Baseline, 3 months, 6 months
  This parameter will allow to describe the clinical evolution of the BMI after application of environmental health measures

SECONDARY OUTCOMES:
Measurement of endocrine disruptors in hair | Change from baseline at 90 days
  Describe the evolution of the amount of endocrine disruptors in hair after the implementation of environmental health measures. from 70 to 100 mg of hair will cut as close as possible to the scalp at the posterior vertex, and stored at room temperature to measure endocrine disruptors such as parabens, phthalates, bisphenols and pesticides.
Tanner scale | Change from baseline at 90 and 180 days
  The Tanner scale is a scale of physical development as children transition into adolescence and then adulthood. The scale defines physical measurements of development based on external primary and secondary sex characteristics.
  Breast:
  Tanner I: no glandular tissue Tanner II: breast bud forms, areola begins to widen Tanner III: breast begins to become more elevated, and extends beyond the borders of the areola, Tanner IV: increased breast sizing and elevation; areola and papilla form a secondary mound projecting from the contour of the surrounding breast Tanner V: breast reaches final adult size
  Pubis hair:
  Tanner I: no pubic hair Tanner II: small amount of long, downy hair Tanner III: hair becomes more coarse and curly, and begins to extend laterally Tanner IV: adult-like hair quality, extending across pubis but sparing medial thighs Tanner V: hair extends to medial surface of the thighs
Bone age determination by X ray | Change from baseline at 90
  Determination of bone age to determine the maturity of the child's skeletal system.
Degree of severity of teeth hypomineralisation | Baseline, 3 months
  The dree of severity is determine according to a scale: 1: <30% of the tooth's enamel surface area visibly disrupted, 2: 31 to 49% of the tooth's enamel surface area visibly disrupted, 3: >50% of the tooth's enamel surface area visibly disrupted
Follicle-stimulating hormone (FSH) level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Estradiol (E2) level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Testosterone Level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
17 hydroxyprogesterone level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Dehydroepiandrosterone sulfate level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Sex Hormone-Binding Globulin level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Thyroid Stimulating Hormone level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
FT4 (Free Thyroxine hormone) level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Androstenedione level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Insulin level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Glycated hemoglobin (HbA1C) level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Insulin-like Growth Factor-1 level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Leptine level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Luteinizing hormone (LH) level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline
Glycemia level | Change from baseline at 90 days and 180 days
  Blood test for determining the evolution of this parameter from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Patricia RANNAUD-BARTAIRE, PhD, Principal Investigator — Hôpital Saint-Vincent de Paul
Locations (2):
- France (2):
  - Cabinet BLM, Lambersart, Hauts-de-France
  - Saint Vincent hospital, Lille, Hauts-de-France

IPD SHARING:
Plan to Share IPD: No